CLINICAL TRIAL: NCT02479542
Title: Randomized Trial Comparing the Negative Pressure Wound Therapy to Standard Gauze Dressings for Acute Wounds in Mbingo Baptist Hospital, Cameroon
Brief Title: Addition of Negative Pressure Wound Therapy to Standard Gauze Dressings for Acute Wounds in a Limited-Resource Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Regulatory issues
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sherry M. Wren MD, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU 34186
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2015-11

CONDITIONS: Wounds and Injuries
Keywords: Negative-Pressure Wound Therapy; Wound Healing; Global Health; Cameroon
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Gauze Dressing (Active Comparator): Patients with wounds that meet eligibility criteria will be randomized, if randomized to the Standard Gauze Dressing Arm, a saline moistened sterile gauze will be packed into the wound with dry gauze and either tape or other means will be used to secure the dressing. The dressing will be changed daily and measured and photodocumented every 72 hours with the Wound Zoom system.
  Interventions: Other: Standard Gauze Dressing
- WiCare NPWT dressing (Experimental): Patients with wounds that meet eligibility criteria will be randomized, if randomized to the WiCare NPWT Dressing Arm, a saline moistened sterile gauze will be packed into the wound and then the WiCare dressing and wound pump will be placed on the wound. The dressing will be changed, measured and photodocumented every 72 hours with the Wound Zoom system.
  Interventions: Device: WiCare NPWT dressing

INTERVENTIONS:
Other: Standard Gauze Dressing — Following consenting of participant, the wound will be photographed with the Wound Zoom imaging system and measured for greatest length, width, and depth. For patients randomized to the control arm, only standard gauze dressings will be applied and changed daily. Wounds with the standard gauze dressings will be photo-documented and measured with the same variables every 72 hours. Wounds and dressing will be evaluated daily for drainage, exudate, presence of infection, and gauze dressings will be changed daily.
  Arms: Standard Gauze Dressing
Device: WiCare NPWT dressing — Following consenting of participant, the wound will be photographed with the Wound Zoom imaging system and measured for greatest length, width, and depth. For patients randomized to the simplified NPWT arm, the standard gauze dressing will be placed then the the WiCare NPWT dressing will be applied. Wounds and WiCare NPWT device will be evaluated daily for drainage, exudate, presence of infection, drainage in pump, integrity of air tight seal. Wounds will be changed by protocol with photo documentation every 72 hours for a total of 18 days or achievement of primary endpoint.
  Arms: WiCare NPWT dressing

SUMMARY:
The worldwide prevalence of open wounds is estimated to be approximately 200 million per year. Negative Pressure Wound Therapy (NPWT), the application of a controlled vacuum to an open wound cavity, has been clinically demonstrated in developed nations to speed the healing time of open wounds by a factor of two or more, and to aid in complete recovery with less scar tissue. Use of NPWT devices has not been feasible in an limited-resource settings due to cost, bulk, and requirement for consistent electricity. This study aims to follow up prior clinical studies that have established the safety and efficacy of simplified NPWT, by assessing changes in wound closure time and wound contraction rate when simplified NPWT is used in a limited-resource setting.

DETAILED DESCRIPTION:
Hypothesis:

Application of WiCare Wound Pump to a standard gauze dressing will result in faster time to definitive wound closure and rate of healing in acute wounds from trauma, infection, or surgery as compared to standard gauze dressing without negative pressure.

Study Design A. Single center prospective trial to be conducted at Mbingo Baptist Hospital (MBH) a multispecialty hospital located in North-West Cameroon that provides complex surgical care.

B. Phase II C. Two arm trial with all patients with eligible wounds offered entrance into Phase II trial D. Blinding: Non E. Indication and patient population: Acute wounds secondary to trauma, infection, or surgical excision in adult patients (>15 year old) F. Sample size: 100 total; based on Schoenfeld's Method to compare two-sample Log-Rank Test with Power of 80%, significance level=5% G. Random Permuted Blocks: Patients will be randomized in blocks of 4 using the following schema Treatment A) WiCare, Treatment B) Standard Dressing: AABB, ABAB, BAAB, BABA, BBAA, and ABBA.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 15 years of age,
* Acute wounds <21 days from any soft tissue traumatic, surgical, or infectious cause.
* Wound size must be either

  1. a minimum of 25 sq cm in cross dimension with a minimum wound depth of 1 cm at the deepest point or
  2. a minimum of 16 sq cm in cross dimension with a minimum depth of 1.5 cm at deepest point.
* Wounds must have been cleaned and debrided of all debris, foreign body contamination (dirt, grass, bone fragments, other debris), necrotic tissue, and pus
* Wound should be considered stable (not evoloving) and ready for dressing changes every 72hours.
* Necrotizing soft tissue infection wounds will only be considered after control of infection through medical and surgical treatment and the wound stable enough for a dressing change every 72 hours.
* Aamputation stump wounds can be included if all other criteria fulfilled.

Exclusion Criteria:

* A wound that would be able to be closed primarily or within 5 days through suture closure, flap rotation or immediate skin graft coverage.
* A wound greater than or equal to 21 cm in either length or width at the initial measurement.
* A wound in the perineum: defined by the pubic bone anteriorly and the anus posteriorly.
* A wound with a visible blood vessel of >3mm.
* The presence of known cancer in the wound.
* Acute burns or burns with skin grafts wound.
* Latex allergy.
* Expected mortality within 30 days of admission from co-exisitng medical or surgical condition.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Time to Wound Closure | 5-19 days following application of dressing
  The effect of simplified negative pressure wound therapy device use on the time to definitive wound closure or time to wound becoming appropriate for discharge for eschar formation.

SECONDARY OUTCOMES:
Rate of Wound Contraction | 5-19 days following application of dressing
  The rate of wound contraction with NPWT for those wounds that do not reach definitive wound closure by study endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry M Wren, MD, Principal Investigator — Stanford University; Brannon Weeks, BA, Principal Investigator — Stanford University

REFERENCES:
- [Background] Saxena V, Hwang CW, Huang S, Eichbaum Q, Ingber D, Orgill DP. Vacuum-assisted closure: microdeformations of wounds and cell proliferation. Plast Reconstr Surg. 2004 Oct;114(5):1086-96; discussion 1097-8. doi: 10.1097/01.prs.0000135330.51408.97. PMID 15457017
- [Background] Borgquist O, Gustafsson L, Ingemansson R, Malmsjo M. Micro- and macromechanical effects on the wound bed of negative pressure wound therapy using gauze and foam. Ann Plast Surg. 2010 Jun;64(6):789-93. doi: 10.1097/SAP.0b013e3181ba578a. PMID 20489409
- [Background] Chariker ME, Gerstle TL, Morrison CS. An algorithmic approach to the use of gauze-based negative-pressure wound therapy as a bridge to closure in pediatric extremity trauma. Plast Reconstr Surg. 2009 May;123(5):1510-1520. doi: 10.1097/PRS.0b013e3181a20563. PMID 19407624
- [Background] Orgill DP, Bayer LR. Update on negative-pressure wound therapy. Plast Reconstr Surg. 2011 Jan;127 Suppl 1:105S-115S. doi: 10.1097/PRS.0b013e318200a427. PMID 21200280
- [Background] Wilkes R, Zhao Y, Kieswetter K, Haridas B. Effects of dressing type on 3D tissue microdeformations during negative pressure wound therapy: a computational study. J Biomech Eng. 2009 Mar;131(3):031012. doi: 10.1115/1.2947358. PMID 19154071
- [Background] Malmsjo M, Ingemansson R, Martin R, Huddleston E. Negative-pressure wound therapy using gauze or open-cell polyurethane foam: similar early effects on pressure transduction and tissue contraction in an experimental porcine wound model. Wound Repair Regen. 2009 Mar-Apr;17(2):200-5. doi: 10.1111/j.1524-475X.2009.00461.x. PMID 19320888
- [Background] Malmsjo M, Ingemansson R, Martin R, Huddleston E. Wound edge microvascular blood flow: effects of negative pressure wound therapy using gauze or polyurethane foam. Ann Plast Surg. 2009 Dec;63(6):676-81. doi: 10.1097/SAP.0b013e31819ae01b. PMID 19887926
- [Background] Dorafshar AH, Franczyk M, Gottlieb LJ, Wroblewski KE, Lohman RF. A prospective randomized trial comparing subatmospheric wound therapy with a sealed gauze dressing and the standard vacuum-assisted closure device. Ann Plast Surg. 2012 Jul;69(1):79-84. doi: 10.1097/SAP.0b013e318221286c. PMID 21712704
- [Background] Dunn R, Hurd T, Chadwick P, Cote J, Cockwill J, Mole T, Smith J. Factors associated with positive outcomes in 131 patients treated with gauze-based negative pressure wound therapy. Int J Surg. 2011;9(3):258-62. doi: 10.1016/j.ijsu.2010.12.005. Epub 2010 Dec 25. PMID 21187174
- [Background] Campbell PE, Smith GS, Smith JM. Retrospective clinical evaluation of gauze-based negative pressure wound therapy. Int Wound J. 2008 Jun;5(2):280-6. doi: 10.1111/j.1742-481X.2008.00485.x. PMID 18494633
- [Background] Jeffery SL. Advanced wound therapies in the management of severe military lower limb trauma: a new perspective. Eplasty. 2009 Jul 21;9:e28. PMID 19696875
- [Background] Lee HJ, Kim JW, Oh CW, Min WK, Shon OJ, Oh JK, Park BC, Ihn JC. Negative pressure wound therapy for soft tissue injuries around the foot and ankle. J Orthop Surg Res. 2009 May 9;4:14. doi: 10.1186/1749-799X-4-14. PMID 19426531
- [Background] Bagheri Nejad S, Allegranzi B, Syed SB, Ellis B, Pittet D. Health-care-associated infection in Africa: a systematic review. Bull World Health Organ. 2011 Oct 1;89(10):757-65. doi: 10.2471/BLT.11.088179. Epub 2011 Jul 20. PMID 22084514
- [Background] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970